CLINICAL TRIAL: NCT00325936
Title: A Multi-Center, Double-Blind, Randomized, Superiority Clinical Study to Compare the Effects of Cilnidipine on Metabolic Syndrome Improvement With Nifedipine GITS in Hypertensive Patients With Metabolic Syndrome (Phase IV) [SLIMS]
Brief Title: The Effects of Cilnidipine on Metabolic Syndrome Improvement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Choi, Jeongeun/Director, Boryung Pharmaceutical Co., Ltd
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNL-MS-01; SLIMS study
Record Dates: First submitted 2006-05-12; First posted 2006-05-15 (Estimated); Last update posted 2008-08-27 (Estimated); Status verified 2008-08

CONDITIONS: Hypertension; Metabolic Syndrome X
Keywords: metabolic syndrome; Hypertension; CCB; cilnidipine
MeSH Terms: conditions — Hypertension; Metabolic Syndrome | interventions — cilnidipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nifedipine (Active Comparator): parrallel design
  Interventions: Drug: Cilnidipine
- Cilnidipine (Experimental)
  Interventions: Drug: Cilnidipine

INTERVENTIONS:
Drug: Cilnidipine — 10~20mg, qd, po for 3 months or 12 months.
  Other Names: Cinalong

SUMMARY:
Abnormalities of glucose, insulin and lipoprotein metabolism are common in patients with hypertension, and these metabolic abnormalities are reported to be related to insulin resistance. Therefore, whenever treating such patients, antihypertensive agents that may have the added effect of improving insulin resistance should be selected. CinalongTM (Cilnidipine) is expected to improve metabolic syndrome as well as insulin resistance by its dual effects on L and N-type calcium (Ca) channels. In this study, the researchers investigate the effects of CinalongTM on insulin resistance and other metabolic related factors.

DETAILED DESCRIPTION:
* Multi-center, randomized, prospective, double blind, active control, parallel study
* Superiority study (Treatment group - Cilnidipine/Control group - Nifedipine)
* Measure the effects of Cinalong(TM) after 3 month and 12 month-application

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, 30-65 years of age having essential hypertension with metabolic syndrome
2. At Screening and Visit 1, blood pressure should be: sitting systolic blood pressure (SiSBP) >=140 mmHg or sitting diastolic blood pressure (SiDBP)>= 90 mmHg and two or more of the following criteria should apply.

   * Abdominal obesity: waist circumference >= 90 cm in men and >= 80 cm in women
   * Hypertriglyceridemia:. >=150 mg/dl (1.695 mmol/l)
   * Low HDL cholesterol: < 40 mg/dl (1.036 mmol/l) in men and < 50 mg/dl (1.295 mmol/l) in women
   * High fasting glucose: >= 110 mg/dl (6.1 mmol/l)

Exclusion Criteria:

1. Secondary hypertension
2. Malignant hypertension

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2005-07; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Homeostasis model assessment of insulin sensitivity (HOMA-IR) | after 3 month and 12 month treatment
Triglyceride/HDL cholesterol ratio | after 3 month and 12 month treatment

SECONDARY OUTCOMES:
Quantitative insulin-sensitivity check index (QUICKI) | after 3 month and 12 month treatment
Resting heart rate | after 3 month and 12 month treatment
Resting norepinephrine | after 3 month and 12 month treatment
Change in abdominal obesity | after 3 month and 12 month treatment
Change in triglyceride | after 3 month and 12 month treatment
Change in cholesterol | after 3 month and 12 month treatment
Decrease in trough SiSBP&SiDBP | after 3 month and 12 month treatment
Change in blood glucose | after 3 month and 12 month treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Bae Park, Ph.D., Study Chair — Cheil General Hospital and Women's Healthcare Center; Sang-hyun Lim, Ph.D., Principal Investigator — Catholic University Holy Family Hospital; Ho-joong Youn, Ph.D., Principal Investigator — Catholic University St Mary's Hospital (Yeouido); Yeong-geun An, Ph.D., Principal Investigator — Chonnam National University Hospital; Dong-su Kim, Ph.D., Principal Investigator — Inje University; Seong-yun Lee, Ph.D., Principal Investigator — Inje University Ilsan Paik Hospital; Heon-sik Park, Ph.D., Principal Investigator — Kyungpook National University Hospital; Ji-dong Seong, Ph.D., Principal Investigator — Samsung Medical Center; In-ho Chae, Ph.D., Principal Investigator — Seoul National University Bundang Hospital; Se-joong Im, Ph.D., Principal Investigator — Youngdong Severance Hospital
Locations (1):
- Cheil general hospital, Seoul, South Korea